CLINICAL TRIAL: NCT05851638
Title: The NIOMI Study: Non-Invasive Lung Oxygen Monitoring of Term Infants
Acronym: NIOMI
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: Tyndall National Institute (Unknown)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Professor, University College Cork
Other Study IDs: 12 MAY 2020/Version 1.0
Record Dates: First submitted 2023-01-25; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Lung Diseases
Keywords: lungs; oxygen; GASMAS; Spectroscopy; neonate
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy term neonates: Inclusion criteria for participant selection are:
  * Healthy infant on postnatal ward.
  * Full term (gestational age ≥37 weeks).
  * Anticipated stay in the hospital > 1 day.
  Exclusion criteria for participant selection are:
  * Parent/guardian unable to/decline to participate in the study.
  * Baby admitted to the Neonatal Unit.
  * Presence of congenital cardiac anomalies (report of antenatal scans from patient electronic record chart).
  Interventions: Device: Lung Oxygen measurement with GASMAS system

INTERVENTIONS:
Device: Lung Oxygen measurement with GASMAS system — A specially designed light source probe (2x2cm size) with 2x incorporated laser sources and a detector probe (2x2cm size) will be attached to the torso of the infant in a total of 10 locations to measure lung oxygen.

SUMMARY:
Infants born prematurely e.g. before 28 weeks of gestational age have a 50% chance of developing neonatal respiratory distress syndrome (NRDS). The management of NRDS is currently driven by information obtained from a sampling of arterial blood, pulse oximetry, and x-ray imaging. On the other hand, these tests carry short and long-term negative outcomes for vulnerable patients. Optical technology has been developed to evaluate lung function non-invasively and without any potential risks for the patients. It is based on Gas in Scattering Media Absorbance Spectroscopy (GASMAS) method, using low-power laser light and a photodetector attached directly to the baby's torso.

DETAILED DESCRIPTION:
The purpose of this observational study is to test a non-invasive, optical system designed to directly measure the oxygen within the lungs of neonates using a GASMAS system (NEOLA-alpha 2, GPX medical). The findings of this study will generate the necessary information that will be used to guide the development of the GASMAS-based systems for future clinical adaptation in preterm infants.

Subjects. The measurements will be performed on full-term (gestational age ≥37 weeks), healthy infants after parental consent has been obtained.

Number of participants to be recruited: 100

Data collection. This will be a prospective study. Relevant data will be collected from maternal and neonatal electronic chart records.

Procedure. A specially designed light source probe (2x2cm size) with 2x incorporated laser sources and a detector probe (2x2cm size) will be attached to the torso of the infant in a total of 10 locations (5 for the left side of the chest and 5 for the right side) to measure lung oxygen.

Locations of the probes. The measurements will be recorded with the detector probe placed in the infant's armpit and the light source probe placed at the locations indicated below:

1. 2nd intercostal space in midclavicular line;
2. 4th intercostal space in midclavicular line (beside the level of nipple);
3. 6th intercostal space in midclavicular line;
4. 1.5 cm below detector probe in midaxillary line;
5. parasternally beside inferior angle of scapula.

Duration. A single optical measurement lasts approximately 2 minutes. The entire measurement session will be aimed to be completed in 30 minutes. Same measurements will be obtained daily until baby will be discharged from the hospital.

Special conditions. This is a painless procedure that should not carry any risks for the baby.

Location. Procedure will be performed in a separate monitoring room on the postnatal ward in Cork University Maternity hospital (CUMH), where parental and infant comfort as well as appropriate handling of technique can be ensured.

Safety measures Materials. The components of the GASMAS system that will be in contact with the infant's skin have been fabricated from non-toxic materials. They were also designed to be as comfortable as possible without any sharp corners or features.

Eye safety. The emission from the light source probe at all wavelengths is weak and diffuse and falls under "Laser Class I" category. Lasers of this category are considered safe and present no hazard to the eye or the skin under direct exposure. There is no need to wear any eye protection for anyone involved in the measurements.

Electrical safety. The system is well shielded and safe to use. Leak currents are tested according to standard 60601. The system has been tested to comply with Radiated Emission Test according to standard EN 55032 Class A.

Mechanical safety. The medical cart is tested to UL/EN/IEC and FCC Part 15 Class A specifications for enhanced patient safety. The medical cart is environmentally clean with RoHS, REACH, WEEE and EU (94/62/EC) packaging compliance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant on the postnatal ward.
* Full-term (gestational age ≥37 weeks).
* Anticipated stay in the hospital > 1 day.

Exclusion Criteria:

* Parent/guardian unable to/declined to participate in the study.
* The baby was admitted to the Neonatal Unit.
* Presence of congenital cardiac anomalies (report of antenatal scans from patient electronic record chart)

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Random parents will be approached on the postnatal ward during working day hours by one of the research team members. The measurements will be performed on full-term, healthy infants after parental consent has been obtained.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of infants in whom at least 1 oxygen measurement was obtained. | 12 months
  The primary outcome will be the percentage of infants in whom at least 1 oxygen measurement was obtained where the signal-to-noise ratio was greater than 3.
Projected concentration in percent meters | 12 months
  Describe the absorption of water vapor and molecular oxygen, by means of projected concentration, presented in percent meters (%m)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Dempsey, Professor, Principal Investigator — University College Cork
Locations (1):
- Cork University Maternity Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided